CLINICAL TRIAL: NCT03078543
Title: A Prospective, Multicentre, Cohort Study Assessing the Safety and Efficacy of the ANTHEM™ PS Total Knee System in Patients Following a Total Knee Arthroplasty
Brief Title: Ten Year Implant Survivorship of the ANTHEM™ PS Total Knee System
Acronym: ANTHEM PS
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-4065-09; OREM-ANTHEM-PMCFU (Other: Smith & Nephew)
Record Dates: First submitted 2017-02-06; First posted 2017-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ANTHEM™ PS Total Knee System implant: The ANTHEM™ PS Total Knee System will demonstrate non-inferiority of 10 year implant survivorship in patients undergoing total knee arthroplasty for osteoarthritis compared to reported literature
  Interventions: Device: ANTHEM™ PS Total Knee System implant

INTERVENTIONS:
Device: ANTHEM™ PS Total Knee System implant — The ANTHEM™ PS Total Knee System is a comprehensive system which allows surgeons to address simple to complex knee arthroplasties. The ANTHEM™ PS Total Knee System consists of the following components:
  * Cobalt-Chrome (Co-Cr) femoral components - Posterior stabilised
  * Titanium primary tibial components
  * Posterior-stabilised ultra-high molecular weight polyethylene (UHMWPE)
  * Polyethylene patella components The resulting product is sufficient to accommodate a wide range of clinical applications.

SUMMARY:
The ANTHEM™PS Total Knee System is being conducted to demonstrate non-inferiority of 10 year implant survivorship in patients undergoing total knee arthroplasty for osteoarthritis compared to reported literature

DETAILED DESCRIPTION:
The ANTHEM PS Study is a prospective, multicentre, cohort study to collect relevant patient reported, clinical, surgical and radiological data from 143 subjects implanted with the ANTHEM™PS Knee System for degenerative joint disease in up to 6 clinical sites globally. Total study duration for study participants will be 10 years with post-operative follow-up visits planned for 6 weeks, 1 year, 2 years, 5 years, 7.5 years and 10 years. The study will evaluate the 10 year implant survivorship and the safety and outcome of the ANTHEM™PS Knee System over 10 years. This is a post-market study of the ANTHEM™PS Total Knee System.

The primary objective of the study is to demonstrate non-inferiority (8% margin) of 10 year implant survivorship of the ANTHEM™PS Total Knee System in patients undergoing total knee arthroplasty for osteoarthritis compared to reported literature.

The secondary objectives of the study are to evaluate shorter and long term safety and outcomes of the ANTHEM™ PS Total Knee System.

* Knee injury and Osteoarthritis Outcomes Score (KOOS)
* 2011 Knee Society Score (2011 KSS)
* EQ-5D - 3L
* Femoral Fit ('Perfect Fit' rate)
* Radiographic Assessment
* Revision for any reason
* Adverse Events (AEs)

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a candidate for primary total knee arthroplasty due to degenerative joint disease
2. Subject is willing to sign and date an EC-approved consent form
3. Subject is male or female between the ages of 18 and 75 years of age
4. Subject plans to be available through ten (10) years post-operative follow-up
5. Subject agrees to follow the study protocol

Exclusion Criteria:

1. Subject would receive the ANTHEM™ Total Knee System on the affected knee as a revision for a previously failed total or unicondylar knee arthroplasty
2. Subject received TKA on the contralateral knee as a revision for a previously failed total or unicondylar knee arthroplasty
3. Subject has a history of patellar fracture, patellectomy, patello-femoral instability
4. Subject has inflammatory arthritis
5. Subject possesses a contralateral or ipsilateral revision hip arthroplasty
6. Subject has ipsilateral hip arthritis resulting in flexion contracture
7. Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the Investigator:

   * Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty
   * Contralateral primary total knee or unicondylar knee arthroplasty
8. Subject has an active infection or sepsis (treated or untreated)
9. Subject has presence of malignant tumor, either primary or metastatic, or benign tumor on leg with the knee to be treated
10. Subject has conditions that may interfere with the TKA survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes mellitus i.e. not under treatment with oral/injectable medications to control blood glucose levels, fibromyalgia, moderate to severe renal insufficiency or neuromuscular disease)
11. Subject has a chronic, contralateral lower extremity condition causing abnormal ambulation, which is not related to the knee (e.g. ankle fusion, ankle arthroplasty, previous hip fracture).
12. Subject is pregnant or plans to become pregnant during the study
13. Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study, including mental illness, mental retardation, drug or alcohol abuse
14. Subject has a BMI>40
15. Subject is enrolled in another investigational drug, biologic, or device study
16. Subject is facing current or impending incarceration
17. Subject has an inadequate bone stock to support the device which would make the procedure unjustifiable, including but not limited to: severe osteopenia/osteoporosis or family history of severe osteoporosis/osteopenia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing primary total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Ten year Anthem knee implant survivorship | Study participants will be followed for 10 years
  The ANTHEM™ Total Knee System will demonstrate non-inferiority of 10 year implant survivorship in patients undergoing total knee arthroplasty for osteoarthritis compared to reported literature

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcomes Score (KOOS) | Participant questionnaire completed at the Baseline timepoint, 6 weeks, 1,2, 5 and 10 years
  Participant Questionnaire to assess the patients opinion about their knee and associated problems.
2011 Knee Society Score (2011 KSS) | Participant questionnaire completed at the Baseline timepoint, 6 weeks, 1,2, 5 and 10 years
  Participant questionnaire including a pre-operative section supplying information relating to the current symptoms, knee function, satisfaction with their pre-operative functional activities, and the expectations they have of the results of the total knee arthroplasty. The surgeon then completes information on objective measures such as joint alignment, instability, motions and symptoms.
EQ-5D-3L | Participant questionnaire completed at the Baseline timepoint, 6 weeks, 1,2, 5, 7.5 and 10 years
  Participant Questionnaire_ The EQ-5D-3L questionnaire is a self-rating evaluation questionnaire made up of health status measurements of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participants also evaluate their overall health status using a visual analogue scale.
Femoral Fit ('Perfect Fit' rate) | Femoral Fit will be measured at surgery, assessed for an estimated 1 hour
  For each individual knee, 'overall femoral component fit' across the combined three femur levels; condylar, junctional and trochlear will be characterised under three classifications:
  1. Perfect Fit: just fit at all three levels or just fit at two levels and underhang at one
  2. Overhang: overhang observed on at least one of the three levels
  3. Underhang: underhang at all three levels or underhang at two and just fit at one
Radiographic Assessments to adequately assess the component position, prosthesis-bone interface, and the knee alignment. | Radiographic assessments to be conducted at Pre-operation timepoint (Baseline), post-operative (Day 1), 6 weeks, 1,2, 5, and 10 years
  The Knee X Rays taken during the course of the study will include Full leg weight-bearing, bilateral anteroposterior (AP), lateral and patellar radiographs. The knee assessments to be made from radiographs will include: Radiographic findings; Component orientation; Radiolucencies; Migration; Osteolysis and Stress shielding.
Revision for any reason | Anytime during the 10 year study period
  Anthem implant revision done for any reason
Adverse Events | Adverse events are collected at any time during the study with formal timepoints being at surgery, 6 weeks, 1,2, 5, 7.5 and 10 years
  All adverse events captured during the entire study period to provide patient safety oversight

CONTACTS AND LOCATIONS:
Overall Officials: Julian Yang, Study Director — Smith & Nephew Medical (Shanghai) Limited
Locations (8):
- Beijing Jishuitan Hospital, Institute of Orthopedics & Traumatology,, Beijing, Beijing Municipality, China
- Italy (2):
  - Instituto Clinico Sant'Ambrogio, Milan, Milan
  - Fatebenefratelli Isola Tiberina Gemelli Hospital - Isle of Rome, Roma
- Westville Hospital, Durban, KwaZulu-Natal, South Africa
- South Korea (3):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam
  - Chonnam National University Hwasun Hospital, Hwasan
  - Severance Hospital, Yonsei University Health System, Seoul
- Siriraj Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No